CLINICAL TRIAL: NCT04202666
Title: The Role of Convex Skin Barrier in Prevention of Peristomy Skin Complication-Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: ConvaTect, Taiwan (Unknown)
Responsible Party: Principal Investigator, Wan-Hsiang Hu, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201901217A3C601
Record Dates: First submitted 2019-11-28; First posted 2019-12-17 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Stoma Colostomy; Stoma Ileostomy
Keywords: peristomy skin complication; convex skin barrier

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- not convex skin barrier (No Intervention): no intervention
- convex skin barrier (Experimental): intervention
  Interventions: Device: convex skin barrier

INTERVENTIONS:
Device: convex skin barrier — Total 300 patients and grouping in 1:1 ratio.(1)peristomy skin complication (30 mins) (2)life quality stomy care (3-5 mins) (3)stomy appliance satisfaction (3-5 mins)
  Arms: convex skin barrier

SUMMARY:
The incidence of peristomy skin complication ranges from 15% to 65%. It is a serious issue and problem for patients care.The type of skin barrier is associated with peristomy skin complication. How to choose suitable skin barrier is important.

ELIGIBILITY:
Inclusion Criteria:

* Age>20
* Receive colostomy or ileostomy
* Agree to join the trial and sign the informed consent form

Exclusion Criteria:

* Liver cirrhosis
* Renal insufficiency
* Severe malnutrition
* Unstable vital sign
* Not suitable after evaluation by Principal Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
peristomy skin complication rate | one month
  peristomy skin complication rate

SECONDARY OUTCOMES:
(2) life quality stomy care questionnaire | one month
  life quality stomy care questionnaire
(3) stomy appliance satisfaction questionnaire | one month
  stomy appliance satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital,Kaohsiung, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Colwell JC, Beitz J. Survey of wound, ostomy and continence (WOC) nurse clinicians on stomal and peristomal complications: a content validation study. J Wound Ostomy Continence Nurs. 2007 Jan-Feb;34(1):57-69. doi: 10.1097/00152192-200701000-00010. PMID 17228209
- [Background] Bosio G, Pisani F, Lucibello L, Fonti A, Scrocca A, Morandell C, Anselmi L, Antonini M, Militello G, Mastronicola D, Gasperini S. A proposal for classifying peristomal skin disorders: results of a multicenter observational study. Ostomy Wound Manage. 2007 Sep;53(9):38-43. PMID 17893429
- [Background] Beitz J, Gerlach M, Ginsburg P, Ho M, McCann E, Schafer V, Scott V, Stallings B, Turnbull G. Content validation of a standardized algorithm for ostomy care. Ostomy Wound Manage. 2010 Oct;56(10):22-38. PMID 21030726
- [Background] Meisner S, Lehur PA, Moran B, Martins L, Jemec GB. Peristomal skin complications are common, expensive, and difficult to manage: a population based cost modeling study. PLoS One. 2012;7(5):e37813. doi: 10.1371/journal.pone.0037813. Epub 2012 May 24. PMID 22679479
- [Background] Hoeflok J, Purnell P. Understanding the role of convex skin barriers in ostomy care. Nursing. 2017 Sep;47(9):51-56. doi: 10.1097/01.NURSE.0000516224.24273.88. No abstract available. PMID 28834934
- [Background] Steinhagen E, Colwell J, Cannon LM. Intestinal Stomas-Postoperative Stoma Care and Peristomal Skin Complications. Clin Colon Rectal Surg. 2017 Jul;30(3):184-192. doi: 10.1055/s-0037-1598159. Epub 2017 May 22. PMID 28684936